CLINICAL TRIAL: NCT02209792
Title: A Randomised, Double-blind, Placebo-controlled, Five* Parallel Groups, Dose Finding Study of BIRB 796 BS (10, 20, 30, and 60 mg*) Administered Twice a Day Orally Over 8 Weeks in Patients With Moderate to Severe Crohn's Disease Followed by a 18 Weeks Treatment Extension in Patients With Clinical Remission or Clinical Response After 8 Weeks Treatment With the Respective Dose of BIRB 796 BS - Extension Phase. * Subsequent to Amendment 4 (Dated 11 Jun 2002) a 60 mg b.i.d. Group Was Included.
Brief Title: Dose Finding Study of BIRB 796 BS in Patients With Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.12
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BIRB 796 BS, low dose (Experimental): 2 x 5 mg b.i.d.
  Interventions: Drug: Placebo; Drug: BIBR 796 BS, 5 mg
- BIRB 796 BS, medium dose 1 (Experimental): 20 mg b.i.d.
  Interventions: Drug: Placebo; Drug: BIBR 796 BS, 20 mg
- BIRB 796 BS, medium dose 2 (Experimental): 2 x 5 mg + 20 mg b.i.d.
  Interventions: Drug: BIBR 796 BS, 5 mg; Drug: BIBR 796 BS, 20 mg
- BIRB 796 BS, high dose (Experimental): 3 x 20 mg b.i.d.
  Interventions: Drug: BIBR 796 BS, 20 mg

INTERVENTIONS:
Drug: Placebo
  Arms: BIRB 796 BS, low dose; BIRB 796 BS, medium dose 1; Placebo
Drug: BIBR 796 BS, 5 mg
  Arms: BIRB 796 BS, low dose; BIRB 796 BS, medium dose 2
Drug: BIBR 796 BS, 20 mg
  Arms: BIRB 796 BS, high dose; BIRB 796 BS, medium dose 1; BIRB 796 BS, medium dose 2

SUMMARY:
The primary objective of this extension study was to obtain long-term safety data for BIRB 796 BS in patients with moderate to severe Crohn's disease after 26 weeks of treatment. Secondary objectives were the evaluation of efficacy of BIRB 796 BS to induce clinical remission and response over 26 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of 18 to 65 years of age
* Provision of written informed consent in accordance with Good Clinical Practice and local legislation prior to any study procedures
* Diagnosis of Crohn's disease documented for at least 6 months. Preferably, inflammatory activity of the bowel should be confirmed by endoscopy within the last 3 months
* Moderate to severe Crohn's disease, CDAI ≥220 to ≤450, at baseline (visit 2)
* Any of the following therapy, provided the respective criteria for dosage, duration and stability were satisfied:

  * Prednisone or other systemic corticosteroids for at least 12 weeks with a stable oral dosage ≤25 mg/d or equivalent for at least two weeks prior to visit 2
  * Budesonide with a stable dose of ≤ 9 mg/d for at least 2 weeks prior to visit 2 (changed by amendment 1, dated 16 January 2002)
  * 5-Aminosalicylic Acid drugs/derivatives, provided they were given for 3 months or more and the dosage was stable for at least 4 weeks prior to visit 2
  * 6-Mercaptopurine or azathioprine, provided they were taken for 6 months or more and the dosage was stable for at least 12 weeks prior to visit 2
  * Methotrexate, provided it was taken for 6 months or more and the dosage was stable and ≤25 mg per week for at least 12 weeks prior to visit 2

The following patients were included in the 18-week treatment extension:

* Patients who received BIRB 796 BS for 8 weeks and reached:

  * Clinical remission (defined as CDAI <150) after 8 weeks or
  * Clinical response (reduction of CDAI ≥70) after 8 weeks
* Patients who were willing to continue with their treatment

Exclusion Criteria:

* Pregnancy (to be excluded at visit 2 by urine β-human chorion-gonadotropin-test in women of childbearing potential) or breast feeding
* Female patients of childbearing potential (not 6 months post-menopausal or surgically sterilised) not using an approved form of birth control (hormonal contraceptives orally or in depot, intrauterine device)
* Patients without signs of inflammation of the bowel in the initial colonoscopy of the substudy
* Patients with colostomy or ileostomy
* Planned or needed surgery during the conduct of the trial due to Crohn's disease or for active gastrointestinal bleeding, peritonitis, intestinal obstruction, or intra-abdominal or pancreatic abscess requiring surgical drainage
* Known or suggested severe fixed symptomatic stenosis of the small or large intestine
* Severe underlying disease in particular of the GI tract (e.g. irritable bowel syndrome, celiac disease, infectious colitis)
* Patients with pathogens or Clostridium difficile toxin detected in the stool culture in the screening period
* Other infectious, ischemic, or immunological diseases with gastrointestinal involvement
* Patients with short bowel syndrome
* Patients who had had a treatment failure with a tumor necrosis factor (TNF)-blocking agent. Treatment failure was defined as not achieving a clinical response (improvement of ≥70 points in CDAI within 4 weeks) in a clinical trial or - in clinical practice -discontinuation of the TNF-blocking agent due to ineffectiveness (changed according to amendment 1, dated 16 January 2002)
* Treatment with cyclosporine A within 12 weeks prior to visit 2
* Last dose given within the specified time period before visit 2 for the following compounds:

  * infliximab (Remicade®): 8 weeks,
  * investigational agent: 4 weeks or 5 half-lives, whichever is longer
* Treatment with anti-inflammatory medication deviating from the criteria for dosage, and stability as provided in the inclusion criteria
* Patients treated with any of the following therapy:

  * antibiotics provided the dosage had not been stable within 2 weeks prior to visit 2;
  * parenteral or elemental diet;
  * intrarectal therapy for Crohn's disease 2 weeks prior to visit 2 (added by amendment 1, dated 16 January 2002)
* Treatment with:

  * Nonsteroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to visit 2;
  * Acetylsalicylic acid >100 mg/d;
  * Paracetamol (acetaminophen) >3 g/day;
  * Drug classified as proton pump inhibitor: 7 days prior to visit 2. This exclusion criterion was deleted after amendment 2 dated 11 June 2002.
  * Drug classified as H2-receptor-blocker or antacid: 2 days prior to visit 2. This exclusion criterion was deleted after amendment 2 dated 11 June 2002.
* Active infection or serious infectious diseases resulting in hospitalisation or requiring systemic anti-infective therapy within 4 weeks before visit 2
* Serologic evidence of active hepatitis B and/or C
* Known HIV-infection
* History of prior tuberculosis infection or suspicion of active infection at screening based on chest X-ray done within 6 months prior to treatment phase
* History of cardiovascular, renal, neurologic, psychiatric, liver, immunologic, or endocrine dysfunction if they were clinically significant. A clinically significant disease was defined as one which, in the opinion of the investigator, may have either put the patient at risk because of participation in the study or as a disease which may have influenced the results of the study or the patient's ability to participate in the study
* Recent history of heart failure (one year or less) or myocardial infarction or patients with any cardiac arrhythmia requiring drug therapy (changed by amendment 1, dated 16 January 2002)
* ECG results outside of the reference range of clinical relevance including, but not limited to QTcB >480 msec, PR interval >240 msec, QRS interval >110 msec
* History of malignant disease in the last 5 years or suspicion of active malignant disease except successfully treated squamous or basal cell carcinoma of the skin and except patients with cervical carcinoma in situ who have had adequate treatment and follow up
* Clinically significant abnormal baseline haematology, blood chemistry or urinalysis if the abnormality defines a disease listed as an exclusion criterion
* Any of the following specific laboratory abnormalities at visit 1:

  * alanine aminotransferase (ALT), aspartate aminotransferase (AST) greater than upper limit of normal range (ULN)
  * Total bilirubin greater than ULN except for patients with documented Gilbert's disease
  * Gamma-glutamyltransferase, alkaline phosphatase or lactate dehydrogenase greater than 1.5 x ULN
  * White blood cell count greater than 1.5 ULN which was not due to Crohn's disease as assessed by the investigator
  * Serum creatinine above 1.5 x ULN
* History of drug or alcohol abuse within the past two years or active drug or alcohol abuse
* Participation in another clinical trial within 4 weeks or 5 half-lives of the respective investigational agent, whichever was longer
* Hypersensitivity to trial drug
* Inability to comply with the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2001-10; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Clinical Remission defined as Crohn's Disease Activity Index (CDAI) < 150 | at week 8

SECONDARY OUTCOMES:
Clinical remission (defined as a CDAI score below 150) | at week 26
Stabilised clinical remission at the end of the main treatment phase | at week 8 and 10
Time to clinical remission | up to 26 weeks
Duration of maintenance of clinical remission | up to 26 weeks
Clinical response (defined as a reduction of CDAI score ≥70) | up to 26 weeks
Time to clinical response | up to 26 weeks
Duration of maintenance of clinical response | up to 26 weeks
Changes from baseline in the CDAI score | up to 26 weeks
Changes from baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) score | up to 26 weeks
Number of patients with 50% fistulae reduction | up to 26 weeks
  defined as an at least 50% reduction from baseline in the number of draining fistulae
Changes from baseline in the number of draining fistulae | up to 26 weeks
Changes from baseline in C-reactive protein (CRP) measurements | up to 26 weeks
Changes from baseline in the daily corticosteroid dose | after week 10
  measured in mg prednisone equivalent
Number of drop-outs due to treatment failure | up to 26 weeks
Number of patients with adverse events | up to 40 weeks
Number of patients with clinically relevant changes in laboratory parameters | up to week 38
Number of patients with relevant findings in electrocardiogram (ECG) | up to 26 weeks
Extended clinical response (defined as a reduction of CDAI score ≥ 100) | week 10 to 26
Time to extended clinical response | week 10 to 26
Duration of maintenance of extended clinical response | week 10 to 26
Changes from baseline in the Crohn's Disease Endoscopic Index of Severity (CDEIS) score | at the end of week 8
  for patients in the endoscopic substudy only
Changes from baseline in the histological scoring of biopsy specimens | at the end of week 8
  for patients in the endoscopic substudy only